CLINICAL TRIAL: NCT01630304
Title: WelTel Retain: Promoting Engagement in Pre-ART HIV Care Through SMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H12-00563; R01MH097558 (NIH)
Record Dates: First submitted 2012-06-25; First posted 2012-06-28 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: HIV
Keywords: telecommunications; Africa; randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WelTel SMS service (Experimental): In addition to standard care, weekly text messages will be delivered to participants randomized to this arm for a one year period. Participants will be requested to respond to the outgoing message "Mambo?" within 48 hours; they may respond that they are doing well (sawa) or that they have a problem (shida). A clinician will call to follow-up with all participants who respond indicating a problem or who do not respond within 48 hours.
  Interventions: Behavioral: WelTel SMS service
- Standard care (No Intervention): This arm will receive standard clinical care.

INTERVENTIONS:
Behavioral: WelTel SMS service — Weekly text message "Mambo?" ("How are you?") to which participants are required to respond either "Shida" (problem) or "Sawa" (OK) within 48 hours. Shida responses and participants who do not respond are called by a clinician.
  Arms: WelTel SMS service

SUMMARY:
The purpose of this study is to determine whether weekly text-messages improve retention in care of HIV-infected individuals who are not yet eligible for antiretroviral therapy (ART).

DETAILED DESCRIPTION:
Patient retention in care is critical to the success of programs funded by the President's Emergency Relief Plan for HIV/AIDS (PEPFAR). High levels of patient retention after first clinical contact contribute to the timely initiation of antiretroviral therapy (ART) and better health outcomes for patients. With the dramatic proliferation of cell phone use in Africa, telecommunications technology offers new opportunities to improve retention using a low-cost, culturally appropriate format. In Kenya (WelTel Kenya1), a weekly short message service (SMS) text message led to improved ART adherence and viral load suppression. This study, WelTel Retain, will evaluate the effect of WelTel on retaining pre-ART patients in care and determine the cost-effectiveness of the intervention. Specific objectives include: 1) determining if the WelTel SMS intervention improves patient retention in the first stage of HIV care; 2) determining whether the WelTel SMS intervention improves 12-month retention; and 3) evaluating the cost-effectiveness of the WelTel SMS intervention. We will fulfil these objectives by conducting a randomized controlled trial at the Kibera Community Health Centre in Nairobi, Kenya. Over one year, HIV positive individuals newly enrolling at the clinic will be recruited and randomly allocated to an intervention or control arm at a 1:1 ratio. Intervention arm participants will receive a weekly SMS 'check-in' to which they will be required to respond within 48 hours. An HIV clinician will follow-up and triage any problems that are identified. The control arm will receive standard of care. Patients will be followed for one year. The WelTel Retain study will contribute critical information on the effectiveness of an mHealth program to engage patients in care during the first year of HIV care. This research has the potential to demonstrate that the WelTel SMS intervention is an effective, feasible retention strategy, which can contribute significantly to the long-term success of PEPFAR-funded programs and towards a sustainable global HIV/AIDS response.

ELIGIBILITY:
Inclusion Criteria:

* evidence of HIV infection
* newly enrolling at the Kibera Community Health Centre
* own or have sufficient access to a cell phone; able to operate a cell phone using simple text-messaging*
* able and willing to provide informed assent/consent to participate *If a participant does not own a phone but has sufficient access to a cell phone (through a partner, relative, etc.), the participant would be able to either 1) use the accessed phone to respond to the text messages themselves; or, if they are unable to text themselves 2) have their partner, relative etc. respond on their behalf.

Exclusion Criteria:

* individuals will be excluded if they do not meet all of the inclusion criteria.
* individuals transferring from other clinics who are already taking ART will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2013-01; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Patient retention in care | 12 months

SECONDARY OUTCOMES:
First ART eligibility assessment | 3 weeks
  Proportion of patients completing 1st eligibility assessment within 3 weeks
Enrolment in HIV care and treatment program | 2 months
  Proportion of patients who complete counselling sessions (3) and are eligible to enrol in the HIV care and treatment program

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Lester, MD, Principal Investigator — University of British Columbia
Locations (1):
- Kibera Community Health Centre, Nairobi, Kenya

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] van der Kop ML, Muhula S, Nagide PI, Thabane L, Gelmon L, Awiti PO, Abunah B, Kyomuhangi LB, Budd MA, Marra C, Patel A, Karanja S, Ojakaa DI, Mills EJ, Ekstrom AM, Lester RT. Effect of an interactive text-messaging service on patient retention during the first year of HIV care in Kenya (WelTel Retain): an open-label, randomised parallel-group study. Lancet Public Health. 2018 Mar;3(3):e143-e152. doi: 10.1016/S2468-2667(17)30239-6. Epub 2018 Jan 30. PMID 29361433
- [Derived] van der Kop ML, Ojakaa DI, Patel A, Thabane L, Kinagwi K, Ekstrom AM, Smillie K, Karanja S, Awiti P, Mills E, Marra C, Kyomuhangi LB, Lester RT. The effect of weekly short message service communication on patient retention in care in the first year after HIV diagnosis: study protocol for a randomised controlled trial (WelTel Retain). BMJ Open. 2013 Jun 20;3(6):e003155. doi: 10.1136/bmjopen-2013-003155. PMID 23794578